CLINICAL TRIAL: NCT03623386
Title: Effect of Mental Imagery Training on Brain Plasticity and Motor Function in Individuals With Parkinson's Disease: A Functional MRI Investigation
Brief Title: Effect of Mental Imagery Training on Brain Plasticity and Motor Function in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000023535; 1K23NS099478-01A1 (NIH)
Record Dates: First submitted 2018-07-27; First posted 2018-08-09 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with PD neurofeedback training (Experimental): Patients will receive neurofeedback training.
  Interventions: Other: PD neurofeedback
- Patients with PD control (Active Comparator): Patients will not receive neurofeedback training.
  Interventions: Other: PD control
- Patients with PD (No Intervention): Patients perform mental imagery (motor and visual aspects combined) in the MRI scanner without neurofeedback training.

INTERVENTIONS:
Other: PD neurofeedback — PD-neurofeedback subjects will practice motor imagery in the MRI scanner and receive neurofeedback on their performance. There will be a total of 10-12 neurofeedback sessions on two separate days. Subjects will continue practicing motor imagery at home every day throughout the study period for 4-6 weeks.
  Arms: Patients with PD neurofeedback training
Other: PD control — PD-control subjects will practice visual imagery (e.g., of scenery, objects, etc., but not of movement) in the MRI scanner and will not receive neurofeedback on their performance. Subjects will continue practicing visual imagery at home every day throughout the study period for 4-6 weeks.
  Arms: Patients with PD control

SUMMARY:
Effect of Mental Imagery Training on Brain Plasticity and Motor Function in Individuals with Parkinson's Disease: A functional MRI investigation.

DETAILED DESCRIPTION:
This project will examine the effect of functional MRI-based neurofeedback on brain plasticity and motor performance in patients with Parkinson's Disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of idiopathic PD defined according to the UK Brain Bank diagnostic criteria and on a stable dopaminergic medication regimen will be included.

Exclusion Criteria:

* Age < 40 years
* Non-English speaking
* Pregnancy
* Breastfeeding
* Excessive alcohol consumption (> 7 drinks per week for women, > 14 drinks per week for men) or substance use
* History of a neurological disorder such as a brain tumor, stroke, central nervous system infection, multiple sclerosis, movement disorder (other than PD), or seizures
* History of schizophrenia, bipolar disorder, attention deficit disorder, or obsessive compulsive disorder
* History of head injury with loss of consciousness
* Metallic surgical implants or traumatically implanted metallic foreign bodies
* Inability to lie flat for about an hour
* Discomfort being in small, enclosed spaces
* Dementia (Montreal Cognitive Assessment score < 21)
* Depression (Beck Depression Inventory-II score > 19)
* Hoehn & Yahr stage > 3 (i.e., able to stand and walk, but not fully independent)
* Focal neurological findings on exam that suggest cerebral pathology other than that associated with parkinsonism
* Motor symptoms that could potentially introduce too much motion artifact in the imaging data (e.g., MDS-UPDRS resting tremor score > 1 in limbs, head/chin tremor, or dyskinesia by history or exam).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sule Tinaz, MD, Phd, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With PD: Patients perform mental imagery (motor and visual aspects combined) in the MRI scanner without neurofeedback training. This was a small pilot arm with no intervention conducted after the completion of the study.
Period: Overall Study
Arm/Group | Patients With PD Neurofeedback Training | Patients With PD Control | Patients With PD
Started | 26 | 28 | 9
Completed | 22 | 22 | 9
Not Completed | 4 | 6 | 0
Not completed — Protocol Violation | 3 | 2 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — COVID-19 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants included in the complete case analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With PD Neurofeedback Training | Patients With PD Control | Patients With PD | Total
Number analyzed (Participants) | 22 | 22 | 9 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.1) | 65.7 (8.8) | 67.4 (6.1) | 66.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 7 | 27
  Male | 12 | 12 | 2 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 22 | 20 | 9 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 22 | 21 | 9 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 9 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in Right Insula-dorsomedial Frontal Cortex Functional Connectivity Strength.
Description: The functional connectivity strength between the subjects' right insula and dorsomedial frontal cortex will be measured at baseline and post-intervention as each group of subjects engages in their respective imagery tasks. Functional connectivity will be measured as the correlation value between the functional MRI signal time courses obtained from these two brain regions.
Time Frame: 4-6 weeks
Population: Complete case analyses and participants in the pilot PD arm did not have these data collected.
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Patients With PD Neurofeedback Training | Patients With PD Control
Number analyzed (Participants) | 22 | 22
percent change from baseline | 93.2 (84.1) | 97.8 (106.6)
Statistical Analysis 1: Comparison: Patients With PD Neurofeedback Training vs Patients With PD Control; Test type: Superiority; p = 0.981, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Resting-state Functional Connectivity Between the Right Insula and Dorsomedial Frontal Cortex.
Description: We will obtain resting-state functional MRI scans from the PD-neurofeedback and PD-control groups at baseline and post-intervention to examine the changes in intrinsic functional connectivity between the right insula and dorsomedial frontal cortex. Functional connectivity will be measured as the correlation value between the functional MRI signal time courses obtained from these two brain regions.
Time Frame: 4-6 weeks
Population: Complete case analyses and participants in the pilot PD arm did not have these data collected.
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Patients With PD Neurofeedback Training | Patients With PD Control
Number analyzed (Participants) | 22 | 22
percent change from baseline | -2.9 (43.7) | 74.2 (58.8)
Statistical Analysis 1: Comparison: Patients With PD Neurofeedback Training vs Patients With PD Control; Test type: Superiority; p = 0.481, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Motor Impairment
Description: We will administer the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III (motor exam) at baseline and post-intervention to the PD-neurofeedback and PD-control groups to measure the change in motor impairment. The MDS-UPDRS part III is a subscale that provides an objective assessment of motor impairment. The scores range between 0-132. Higher scores indicate more severe impairment.
Time Frame: Baseline and 4-6 weeks
Population: Complete case analyses and participants in the pilot PD arm did not have these data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With PD Neurofeedback Training | Patients With PD Control
Number analyzed (Participants) | 22 | 22
score on a scale
  Pre | 32.3 (8.1) | 34.5 (9.6)
  Post | 31.3 (9.8) | 35.1 (10.8)
Statistical Analysis 1: Comparison: Patients With PD Neurofeedback Training vs Patients With PD Control; Testing for main effects (group), time effect and the interaction of group and time; Test type: Superiority; p > 0.05, ANOVA

4. Primary Outcome: Change in Motor Function
Description: We will administer standard motor function tests (e.g., timed up and go, 5 times sit-to-stand, 360-degree turn) at baseline and post-intervention to the PD-neurofeedback and PD-control groups to measure the change in motor function. The performance score on these tests is the time to complete the motor tasks. Shorter time indicates better performance. The motor function tests measure movement speed. Timed up and go test measures (seconds) how fast one can stand up from a chair, walk 3 meters, turn, walk back to the chair and sit down again. Five times sit-to-stand test measures (seconds) how fast one can stand up from a chair with arms crossed across the chest and sit back again 5 times in a row. 360-degree turn test measures (seconds) how fast one can turn around their own axis clockwise and counterclockwise. The composite motor function score is the sum of the durations (seconds) of all three tests.
Time Frame: Baseline and 4-6 weeks
Population: Complete case analyses and participants in the pilot PD arm did not have these data collected.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Patients With PD Neurofeedback Training | Patients With PD Control
Number analyzed (Participants) | 22 | 22
seconds
  Pre | 23.7 (4.7) | 24.4 (4.9)
  Post | 22.3 (5.1) | 24.1 (5.2)
Statistical Analysis 1: Comparison: Patients With PD Neurofeedback Training vs Patients With PD Control; Testing for main effects (group), time effect and the interaction of group and time; Test type: Superiority; p = 0.026, ANOVA — p value reflects the effect of time

5. Other Pre Specified Outcome: Task-based Functional Connectivity
Description: In a group of PD patients who will not receive any intervention, we will collect functional MRI data during a mental imagery task with both motor and visual imagery components to investigate the functional connectivity between the motor and visual networks.
Time Frame: 1 day
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Patients With PD Neurofeedback Training | Patients With PD Control | Patients With PD
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28 | 0/9
Other Adverse Events (participants affected / at risk) | 0/26 | 0/28 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03623386/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03623386/ICF_001.pdf